CLINICAL TRIAL: NCT01550406
Title: Use of Polyethylene Glycolic Acid or Tachocomb to Prevent Pancreatic Fistula Following Distal Pancreatectomy: Prospective Multicenter Randomized Study
Brief Title: Use of Polyethylene Glycolic Acid or Tachocomb to Prevent Pancreatic Fistula Following Distal Pancreatectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PFDP-2011
Record Dates: First submitted 2011-11-21; First posted 2012-03-12 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Pancreatic Fistula
Keywords: Pancreatic fistula; distal Pancreatectomy
MeSH Terms: conditions — Pancreatic Fistula

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tachocomb (Active Comparator): Tachocomb will be applicated on the cut surface of distal pancreatectomy
  Interventions: Device: Tachocomb
- PGA (Active Comparator): PGA will be applicated on the cut surface of distal pancreatectomy
  Interventions: Device: Polyglycolic acid (PGA) (Neoveil)
- Control (No Intervention): No mesh will be applicated on the cut surface of distal pancreatectomy

INTERVENTIONS:
Device: Tachocomb — A kind of Mesh:
  ready-to-use hemostatic agent consisting of a collagen sheet coated on one side with human fibrinogen, bovine thrombin, and bovine aprotinin
  Arms: Tachocomb
Device: Polyglycolic acid (PGA) (Neoveil) — Polyglycolide or Polyglycolic acid (PGA) is a biodegradable, thermoplastic polymer and the simplest linear, aliphatic polyester.
  Other Names: Neoveil
  Arms: PGA

SUMMARY:
To date, there has been many methods suggested to reduce pancreatic fistula. But there are no evidence of superiority to the other methods. This study is a multicenter prospective randomized phase III study of use of Tachocomb or Polyethylene Glycolic Acid (PGA) to prevent of pancreatic fistula after distal pancreatectomy.

DETAILED DESCRIPTION:
Distal pancreatectomy has been called to by various names such as, left-sided pancreatectomy, distal partial pancreatectomy. It is difficult to define which part of the pancreas as distal in exactly, but typically the superior mesenteric vein (SMV) and splenic vein, come to meet portal vein to form the area that covers the pancreas, neck actually based on a relatively thin pancreatic resection area, if left to its distal pancreatic resection is generally defined as that.

Indication of distal pancreatectomy in Western countries have been trauma (16%), pancreas cancer (18%), neuroendocrine tumors (14%), chronic pancreatitis (24%), other benign disease (22%) and in Korea, in contrast, disease caused by inflammatory process such as chronic pancreatitis has had relatively low incidence. But the rate of combined resection of distal pancreas at the time of gastric surgery was relatively high.

Definitions and names of pancreatic fistula have been reported differently in each center. Heidelberg and Johns Hopkins groups defined pancreatic fistula as drain amylase levels more than three times of normal serum value , and with more than 50mL during 24 hours after postoperative 10 days. German and Italian groups defined that as drain amylase levels more than three times of normal serum value, and with more than 10mL during 24 hours after postoperative 3-4 days. Japanese group defined pancreatic fistula as drain amylase levels more than three times of normal serum value, and with persistent drainage after postoperative 7 days. Lowy et al defined clinically significant pancreatic fistula as 38℃ or more of fever and leukocytosis (> 10,000 cells/mm3), and sepsis associated or necessity of drainage of abdominal fluid.

To adjust this various criteria, International Study Group Pancreatic Fistula (ISGPF) 2005 defined pancreatic fistula as drain amylase levels more than three times of normal serum value at the time of postoperative 3 days, and divided severity by 3 category with A to C in accordance with clinical course.

As followed previous studies, pancreatic fistula has been one of major postoperative complications (13-64%), which is leading cause of intra-abdominal infections, abscesses, septicemia, wound infection, postoperative bleeding, and malnutrition Risk factors related pancreas fistula have been presented as a disease- associated factors (pancreatic hardness, pathological findings, diameter of main p- duct, and the thickness of pancreas resection area), surgery-related factors (method of pancreas resection, intraoperative blood loss, operative time, blood transfusion during surgery), patient-related factors (age, sex, race, comorbidity) and the experience of surgeon, etc.

Based on experience and observation of the above listed risk factors for pancreatic fistula, there has been rarely reported that the incidence of pancreatic fistula was markedly reduced by some kind of methods.

As mentioned above, one of the risk factors of pancreatic fistula is operative method or technique. To date, there has been many methods suggested to reduce pancreatic fistula. For example, as dealing with pancreas cut surface, there has been several methods, such as, hand-sewn suture techniques, stapled closure, the use of fibrin glue, the use of mesh. But there are few evidence of superiority to the other methods.

Recent retrospective studies suggested the usefulness of mesh that the incidence of pancreatic fistula with mesh (5.6-27%) was lower than without mesh (38.9~42.0%).

There are two kind of mesh to use surgical fields, that are PGA and tachocomb. Among that, the methods with PGA has been reported in a few retrospective study. Moreover, there are no report about the effectiveness with Tachocomb.

The objective of this prospective multicenter randomized study is to clarify the proper method to reduce pancreatic fistula by PGA or tachocomb.

ELIGIBILITY:
Inclusion Criteria:

* Expected survival time more than 12 months
* Patients with at least one of the following pathologic diseases scheduled for elective resection

  * Resectable malignancies of the pancreatic body/ tail
  * Resectable pre-malignant lesions of the pancreatic body/ tail
  * Resectable benign lesion of the pancreatic body/ tail

Exclusion Criteria:

* Current immunosuppressive therapy
* Pancreatic atrophy or calcification due to severe pancreatitis
* Chemotherapy or radiotherapy before operation
* Severe psychiatric or neurologic diseases
* Drug- and/or alcohol-abuse according to local standards
* Participation in another intervention trial with interference of a primary or secondary endpoint of this study
* Inability to follow the instructions given by the investigator
* Lack of compliance

Ages: 20 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-11; Primary Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
The rate of pancreatic fistula between groups | postoperative 3rd day
  Pancreatic fistula was defined by criterion of ISGPF, Output through an operatively placed drain or a subsequently placed percutaneous drain, of any measurable volume of drain fluid on or after postoperative day 3, with an amylase content greater than three times the upper normal serum value

SECONDARY OUTCOMES:
Surgery-related risk factor | intraoperative time
  Amount of intraoperative bleeding, blood transfusion, operative time, operative method with open, laparoscopic, or robotic surgery
disease- associated factors | intraoperative time, within 1 day after operation
  pancreatic hardness, pathological findings, diameter of main p- duct, and the thickness of pancreas resection area
patient-related risk factors analysis | 1 week before the operation
  age, sex, race, comorbidity

CONTACTS AND LOCATIONS:
Overall Officials: Jin- Young Jang, M.D., Study Chair — Seoul National University Hospital
Locations (5):
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam, Bundang-gu
  - Department of Surgery, Seoul National University College of Medicine, Seoul
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul

REFERENCES:
- [Derived] Jang JY, Shin YC, Han Y, Park JS, Han HS, Hwang HK, Yoon DS, Kim JK, Yoon YS, Hwang DW, Kang CM, Lee WJ, Heo JS, Kang MJ, Chang YR, Chang J, Jung W, Kim SW. Effect of Polyglycolic Acid Mesh for Prevention of Pancreatic Fistula Following Distal Pancreatectomy: A Randomized Clinical Trial. JAMA Surg. 2017 Feb 1;152(2):150-155. doi: 10.1001/jamasurg.2016.3644. PMID 27784046
- [Derived] Park JS, Lee DH, Jang JY, Han Y, Yoon DS, Kim JK, Han HS, Yoon Y, Hwang D, Kang CM, Hwang HK, Lee WJ, Heo J, Chang YR, Kang MJ, Shin YC, Chang J, Kim H, Jung W, Kim SW. Use of TachoSil((R)) patches to prevent pancreatic leaks after distal pancreatectomy: a prospective, multicenter, randomized controlled study. J Hepatobiliary Pancreat Sci. 2016 Feb;23(2):110-7. doi: 10.1002/jhbp.310. Epub 2016 Jan 19. PMID 26681272